CLINICAL TRIAL: NCT01608971
Title: The Effects of Heparin Level Based Versus Weight Based Protamine Dosing on Protamine Demand, Markers of Haemostasis, Blood Product Utilization and Perioperative Blood Loss in Patients Undergoing Extended Cardiac Surgery Cardiac Surgery
Brief Title: Protamine in Cardiac Surgery and Haemostasis
Acronym: PROTT
Status: Completed | Type: Observational
Sponsor: Heart and Diabetes Center North-Rhine Westfalia (Other)
Responsible Party: Principal Investigator, Andreas Koster, Senior anaestetist, Heart and Diabetes Center North-Rhine Westfalia
Other Study IDs: 007
Record Dates: First submitted 2012-05-29; First posted 2012-05-31 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-02

CONDITIONS: Bleeding; Hemorrhage
Keywords: Protamine; heparin level; haemostasis; thromboelastometry; cardiac surgery; Patients undergoing cardiac surgery
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Weight based protamine group: In this group the dose of protamine is calculated by the weight of the patients (400 IU/kg)
- Heparin level based protamine group: In this group the protamine dose will be calculated 1:1 according to the heparin level measured after termination of cardiopulmonary bypass.

SUMMARY:
Protamine is used after Cardiopulmonary Bypass (CPB) to reverse the anticoagulant effects of heparin and restore coagulation. Convincing evidence from in-vitro and in-vivo studies suggest that an overdose of protamine has anticoagulant effects which might lead to bleeding complications. Heparin levels usually decrease during cardiac surgery with CPB. Therefore, a protamine regimen based on the initial heparin dose before CPB might lead to overdose of protamine. In contrast, a protamine regimen based on the actual heparin concentration may avoid this condition. The investigators compare both regimens of protamine dosing in patients undergoing complex surgery with CPB and assess its effect on the amount of protamine given, markers of the coagulation system, utilization of blood products and perioperative blood loss.

DETAILED DESCRIPTION:
Before induction of anesthesia, patients are randomized to the two different dosing regimen for protamine. Both, the anesthetist and the surgeon were blinded regarding the grouping of the patients.

Anesthesia and CPB

Anesthesia is performed as a balanced anesthesia with a bolus of fentanyl, etomidate, pancuronium-bromide followed by a continuous infusion of remifentanil and vaporization of sevoflurane. Additionally, in all patients a continuous infusion of 0.25 µg/kg/min milrinone will be started after induction of anesthesia. Further inotropic or vasoactive agents (Dobutamine 3-5 µg/kg/min; epinephrine 0.05-0.2 µg(kg/min, norepinephrine 0.05-0.2 µg/kg/min) will be only given when a target cardiac index of < 2.2 l/m² BSA and mean arterial pressure of >70 mmHg is not achieved with this therapy.

In order to compensate the degree of hemodilution due to differences in weight, in patients with a body surface area (BSA) of <1.8 m², a CPB system with a priming volume of 1100 ml will be used while in patients with a BSA of >1.8m² a system with a priming volume of 1500 ml was employed. CBP will be performed with open non-coated CPB circuits in mild hypothermia with a core temperature of 32-34°C. Cardioplegia will be achieved using warm blood cardioplegia according to Calafiore.

All patients receive tranexamic acid (TA) with a bolus of 1 g to the patient, 0.5 g added to the CPB volume and a continuous infusion of 0.2 g/hour during CPB.

Heparin and Protamine Management

Heparin will be given with a bolus of 400 IU/kg to achieve a target celite ACT (Actalyke ACT, Helena Lab. Beaumont, TX USA) value of >450 seconds. If this target is not reached, additional boluses of 1/3 rd of the first dose will be given until prolongation to the target value is achieved. Additional 10.000 units of heparin will be given into the priming volume of the CPB circuit.

Heparin concentrations were measured five minutes after beginning of CPB using the white (range 3.4-6.8 IU/ml heparin) heparin protamine titration (HPT) cartridge of the Hepcon HMS Plus™ device (Medtronic INC, Minneapolis, Min, USA) and shortly after termination of CPB using the golden HPT cartridge (range 2.0 - 5.4 IU/ml heparin).

The total protamine dose consists of 100 ml. Of this 80 ml will be given as a short infusion over 10 min. directly after termination of CPB. The remaining 20 ml will be given when the residual CPB blood is re-infused into the patient after arterial decannulation, which will be performed 10-15 minutes after weaning from CPB.

In the weight based protamine group (Group 1, the total amount of protamine will be calculated 1:1 according to the initial heparin dose necessary to achieve the target ACT of >450 sec. In the heparin level based group, the total protamine amount will be calculated 1:1 according to the actual heparin level measured after termination of CPB with the use of Hepcon HMS Plus™ device.

Coagulation Tests

Fifteen minutes after infusion of protamine, the INTEM, FIBTEM and HEPTEM test will be performed on the ROTEM thromboelastometry system (TEM International GmbH, Munich Germany). In all tests, the coagulation time (CT) reflects the period until clot formation starts; the clot formation time (CFT) reflects the period until a clot strength of 20 mm is achieved and the maximal clot firmness MCF)reflects the maximal clot strength. In the INTEM test the intrinsic coagulation pathway is activated.

Transfusion triggers

During CPB the critical hemoglobin (Hb) triggering transfusion of packed red blood cells (PRBC) is defined at 8 g/dl. After CPB, in patients with a CI >2.2 l/m² the critical value is at >8-9 g/dl, while in patients needing further medical support with dobutamine/epinephrine or norepinephrine the minimum target was defined at >9-10 g/dl.

In patients with diffuse bleeding after protamine administration, therapy with fresh frozen plasma (FFP), prothrombin complex concentrate (Beriplex, CSL Behring, Marburg, Ger) , fibrinogen concentrate (Haemocomplettan P®, CSL Behring, Marburg, Germany) and single donor aphaeresis platelet concentrates will be based on the results of the ROTEM analysis. However, these blood products will only be given when diffuse microvascular bleeding is observed in the operation field.

In case of a moderate prolongation of the CT (240-360 sec) in the INTEM test (and comparable result in the HEPTEM test) 3-4 units of FFP will be transfused. If bleeding persists, additional 3-4 units of FFP or in case of a prolongation of the CT>360 sec. 2000-4000 IU of prothrombin complex concentrate will be given.In case of an MCF < 45 mm to platelet concentrates will be transfused.

ELIGIBILITY:
Inclusion Criteria:

* Primary surgery
* Preoperative hemoglobin value < 12 g/l
* Preoperative platelet count < 200 c/µl
* Patients with a body weight < 50 kg
* No known defect of the coagulation system
* Normal pre-operative ROTEM values of the INTEM and FIBTEM
* Patients with unimpaired renal function (creatinine clearance < 30 ml/kg/min)

Exclusion Criteria:

* <18 years
* No informed consent
* Re-do surgery
* Known defect of the coagulation system
* Renal impairment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing complex cardiac surgery using cardiopulmonary bypass with mitral valve repair/replacement and 2-4 coronary artery bypass grafting including the left thoracic artery
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Koster, MD, Principal Investigator — Heart & Diabetes Center NRW, Ruhr University Bochum, 32545 Bad Oeynhausen, Germany
Locations (1):
- Heart & Diabetes Center NRW, Bad Oeynhausen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Koster A, Borgermann J, Gummert J, Rudloff M, Zittermann A, Schirmer U. Protamine overdose and its impact on coagulation, bleeding, and transfusions after cardiopulmonary bypass: results of a randomized double-blind controlled pilot study. Clin Appl Thromb Hemost. 2014 Apr;20(3):290-5. doi: 10.1177/1076029613484085. Epub 2013 Apr 4. PMID 23564056

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Heparin Level Based Protamine Group | Weight Based Protamine Group
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Weight Based Protamine Group | Heparin Level Based Protamine Group | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 11 | 12 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 10 | 6 | 16
Region of Enrollment [Number; unit: participants]
  Germany | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: INTEM HEPTEM and FIBTEM Test of the ROTEM Coagulation Analyzer
Description: The Intem test of the ROTEM analyzer evaluates the response of the heamostatic system to activation of the intrinsic coagulation system. The following parameters of the INTEM test will be analyzed. CT [seconds](coagulation time), CFT [seconds] (clot formation time) and the CT [seconds] of the HEPTEM test which is non sensitive for residual heparine.
Time Frame: Tests will be measured 15 minutes after Protamine infusion
Population: Rotem INTEM CT, CFT, MCF and FIBTEM MCF and Heptem CT
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Heparin Level Based Protamine Group | Weight Based Protamine Group
Number analyzed (Participants) | 15 | 15
seconds
  CFT Intem | 98 [78 to 131] | 117 [103 to 170]
  CT Intem | 178 [163 to 199] | 253 [202 to 371]
  CT Heptem | 185 [169 to 201] | 267 [209 to 333]

2. Secondary Outcome: Transfusion of Blood Products and Coagulation Factors
Description: The transfusion of blood products and coagulation factors will be assesed from protamine administration until 12 hours postoperatively .
Time Frame: From protamine administration until 12 h after surgery
Population: Transfusion of RBC
Measure: Number; unit: percentage of patients transfused
Arm/Group | Weight Based Protamine Group | Heparin Level Based Protamine Group
Number analyzed (Participants) | 15 | 15
percentage of patients transfused
  RBC transfusion | 76.7 | 80
  PCC transfusion | 20 | 60
  FFP transfusiom | 20 | 60
  RDPC transfusion | 7 | 15
  Fibrinogen transfusion | 33.3 | 20

3. Secondary Outcome: 12 h Postoperative Blood Loss
Description: The intra and postoperative blood loss from the time point of protamine administration until 12 hours postoperatively will be analyzed.
Time Frame: 15 min after protamine administration until 12 hours postoperatively
Measure: Median (Inter-Quartile Range); unit: ml/12 hour
Arm/Group | Weight Based Protamine Group | Heparin Level Based Protamine Group
Number analyzed (Participants) | 15 | 15
ml/12 hour | 620 [600 to 700] | 723 [600 to 850]

4. Primary Outcome: Rotem MCF Fibtem and MCF Intem
Description: The following parameters of the INTEM test will be analyzed: MCF [mm] (maximum clot firmness) which correlates with the platelet count. Furthermore, the MCF [mm] of the FIBTEM test will be analyzed, which correlates with the fibrinogen concentration.
Time Frame: 15 Minutes after protamine infusion
Population: Patients of both groups
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Heparin Level Based Protamine Group | Weight Based Protamine Group
Number analyzed (Participants) | 15 | 15
mm
  MCF Intem | 55 [51 to 60] | 57 [53 to 63]
  MCF Fibtem | 9 [7 to 14] | 13 [10 to 15]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Heparin Level Based Protamine Group | Weight Based Protamine Group
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Heparin Level Based Protamine Group (N=15) | Weight Based Protamine Group (N=15)
Excessive bleeding (Blood and lymphatic system disorders) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
small study cohort

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes